CLINICAL TRIAL: NCT07040605
Title: Effect of Deep Cervical Flexor Muscle Training and Sensorimotor Training in Patient With Chronic Mechanical Neck Pain
Brief Title: Deep Cervical Flexor and Sensorimotor Training for Chronic Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Neelain University (Other)
Responsible Party: Principal Investigator, Halla Taj Elsir Ahmed, lecturer of orthopaedic physical therapy, faculty of physical therapy, Al-Neelain University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005888
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Mechanical Neck Pain
Keywords: mechanical neck pain; sensorimotor training; Deep cervical flexors muscles

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core stability exercise and proprioception training (Experimental): Participants in the experimental group will receive a structured four-week physiotherapy intervention consisting of conventional physical therapy treatment combined with deep cervical flexor muscle training and proprioception (sensorimotor) training.
  Interventions: Other: Deep cervical flexors muscle training and sensorimotor training
- conventional physical therapy exercise (Active Comparator): . Conventional physiotherapy will include stretching exercises targeting the sternocleidomastoid, upper trapezius, levator scapulae, scalene, Rhomboids and pectoralis muscles, performed in three repetitions, holding each stretch for thirty seconds, strengthening exercises will be provided Isometrically for the cervical flexors, extensors and at sides using a prescription of three sets of ten repetitions with a ten-second hold and two minutes of rest between sets.
  TENS for 15 min. hot back for 15 min.
  Interventions: Other: conventional physical therapy exercise

INTERVENTIONS:
Other: Deep cervical flexors muscle training and sensorimotor training — deep cervical flexor muscle training will be performed according to the protocol of Jull and Falla using a pressure biofeedback unit. Participants will be positioned in a supine crook-lying posture with the neck in a neutral position, and the air bag of the pressure biofeedback unit will be placed beneath the cervical lordosis and inflated to a baseline of 20 mmHg. Patients will be instructed to perform a gentle nodding action, increasing the pressure by 2 mmHg increments up to 30 mmHg. Each increment will be held for ten seconds, repeated in three sets of ten repetitions, with a two-minute rest between sets. To enhance activation of the deep flexors, patients will be instructed to keep their mouth open during the exercise.
  Proprioception training will include head relocation practice, oculomotor exercises, and eye-head coordination exercises.
  Arms: core stability exercise and proprioception training
Other: conventional physical therapy exercise — will include stretching exercises targeting the sternocleidomastoid, upper trapezius, levator scapulae, scalene, Rhomboids and pectoralis muscles, performed in three repetitions, holding each stretch for thirty seconds, strengthening exercises will be provided Isometrically for the cervical flexors, extensors and at sides using a prescription of three sets of ten repetitions with a ten-second hold and two minutes of rest between sets.
  TENS and Hot back.
  Arms: conventional physical therapy exercise

SUMMARY:
This randomized controlled trial aims to investigate the effectiveness of deep cervical flexor muscle training combined with sensorimotor (proprioception) training in patients with chronic mechanical neck pain. The study will be conducted in outpatient clinic of the faculty of physical therapy- Cairo University, involving 60 participants aged 20-40 years with neck pain persisting for more than three months. Participants will be randomly allocated into an experimental group receiving conventional physical therapy plus deep flexor and sensorimotor training, and a control group receiving conventional treatment alone. Outcome measures will include pain intensity, craniovertebral angle (CVA), cervical range of motion (ROM), segmental mobility, neuromotor control, proprioception (head repositioning accuracy), and respiratory function (FEV1 and PEF). Assessments will be performed at baseline and after four weeks of intervention. The study seeks to provide evidence-based recommendations for physiotherapy management of mechanical neck pain, particularly addressing the gaps in literature within the regional context.

DETAILED DESCRIPTION:
Participants in the experimental group will receive a structured four-week physiotherapy intervention consisting of conventional physical therapy treatment combined with deep cervical flexor muscle training and proprioception (sensorimotor) training. All participants will attend three supervised sessions per week, with each session lasting approximately 45-60 minutes. Conventional physiotherapy will include stretching exercises targeting the sternocleidomastoid, upper trapezius, levator scapulae, scalene, Rhomboids and pectoralis muscles, performed in three repetitions, holding each stretch for thirty seconds, strengthening exercises will be provided Isometrically for the cervical flexors, extensors and at sides using a prescription of three sets of ten repetitions with a ten-second hold and two minutes of rest between sets.

In addition, deep cervical flexor muscle training will be performed according to the protocol of Jull and Falla using a pressure biofeedback unit. Participants will be positioned in a supine crook-lying posture with the neck in a neutral position, and the air bag of the pressure biofeedback unit will be placed beneath the cervical lordosis and inflated to a baseline of 20 mmHg. Patients will be instructed to perform a gentle nodding action, increasing the pressure by 2 mmHg increments up to 30 mmHg. Each increment will be held for ten seconds, repeated in three sets of ten repetitions, with a two-minute rest between sets. To enhance activation of the deep flexors, patients will be instructed to keep their mouth open during the exercise.

Proprioception training will include head relocation practice, oculomotor exercises, and eye-head coordination exercises. Head relocation exercises will be conducted using a laser pointer attached to a helmet, with participants practicing relocating their head to a neutral position or predetermined positions, initially with eyes open using visual feedback and later progressing to eyes closed. Oculomotor exercises will begin with eye movements while keeping the head stationary, progressing to combined head and eye movements following visual targets. Eye-head coordination exercises will involve moving the eyes and head to the same side, followed by movements where the eyes lead and the head follows, and eventually progressing to eyes and head moving in opposite directions. Exercises will be progressed by increasing speed, range, and target difficulty. This proprioceptive training will also be performed three times per week for four weeks.

The control group will receive the conventional physical therapy program alone, without the additional deep cervical flexor or proprioception training components. Outcome measures for both groups will be assessed at baseline and after four weeks, including pain intensity using the Numeric Pain Rating Scale (NPRS), craniovertebral angle measured by the APECS mobile application, cervical range of motion via Digital Inclinometer, Segmental mobility using spinal mouse, neuromotor control using the Craniocervical Flexion Test with a pressure biofeedback unit, proprioception assessed through head repositioning accuracy tests, and respiratory function parameters (FEV1 and peak expiratory flow) measured with the spirometer.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 20-40 years.
* participant having neck pain report more than 4 in NPRS, and at least within the last three months known as chronic pain.
* participant with CVA more than 45 degrees and less than 50.
* Participant with poor cervical muscle endurance.

Exclusion Criteria:

* Participant with acute neck pain (less than three month).
* Participant with radiated neck pain.
* Participant who undergone recent surgeries within the thoracic, shoulder girdle, and cervical spine regions.
* Participants who were already undergoing treatment for neck pain.
* Participant with fixed spinal deformity.
* Pregnant women.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity Score on the Numeric Pain Rating Scale (NPRS) from Baseline to 4 Weeks | 4 weeks
  which will be measured using the Numeric Pain Rating Scale (NPRS), a validated 11-point scale ranging from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Change in Cervical Range of Motion (ROM) in Degrees Measured by Digital Inclinometer from Baseline to 4 Weeks | 4 weeks
  Flexion, Extension and Rotation range will be assessed using the Digital Inclinometer,
Change in Neuromotor Control of the Deep Cervical Flexor Muscles Assessed by Craniocervical Flexion Test (CCFT) from Baseline to 4 Weeks | 4 weeks
  will be evaluated using the Craniocervical Flexion Test (CCFT) with a pressure biofeedback unit (PBU),
Change in Craniovertebral Angle (CVA) Measured by AI Posture Evaluation and Correction System (APECS) from Baseline to 4 Weeks | 4 weeks
  will be used as a key postural assessment parameter, measured via the AI Posture Evaluation and Correction System (APECS) mobile application, which provides reliable digital posture analysis using lateral photographic images to quantify forward head posture.
Change in Cervical Proprioceptive Function Assessed by Head Repositioning Accuracy (HRA) Test in centimetre from Baseline to 4 Weeks | 4 weeks
  will be evaluated through the Head Repositioning Accuracy (HRA) Test,
Change in Respiratory Function Parameters (FEV1 and PEF) Measured by Spirometer from Baseline to 4 Weeks | 4 weeks
  will be assessed by measuring forced expiratory volume in the first second (FEV1) and peak expiratory flow (PEF) using the spirometer

CONTACTS AND LOCATIONS:
Overall Officials: Khaled A Ayad, Professor, Study Chair — Cairo University; Karima A Mohamed, PhD, Study Director — Cairo University
Locations (1):
- Out-patient clinic- Faculty of physical therapy, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study result
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after publication
Access Criteria: study protocol